CLINICAL TRIAL: NCT04650243
Title: Clinical Research of Tapering Ursodeoxycholic Acid in Primary Biliary Cholangitis Patients With A Complete Response
Brief Title: Clinical Research of Tapering UDCA in PBC Patients With a Complete Response
Acronym: UDCA PBC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-2237
Record Dates: First submitted 2020-04-27; First posted 2020-12-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: Primary Biliary Cholangitis
Keywords: ursodeoxycholic acid; reducing medication regimen
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: In our study, the 90 recruited PBC patients with a complete response will be distributed randomly into two experimental groups and one control group. The two experimental groups will receive reduced dosage of UDCA at 10mg/Kg and 5mg/Kg respectively, while the control group will receive standard 13-15mg/Kg UDCA. The effect of therapy will be evaluated every three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 10mg/Kg UDCA (Experimental): Patients will receive a reduced dosage of 10mg/Kg UDCA orally everyday.
  Interventions: Drug: ursodeoxycholic acid
- 5mg/Kg UDCA (Experimental): Patients will receive a reduced dosage of 5mg/Kg UDCA orally everyday.
  Interventions: Drug: ursodeoxycholic acid
- standard 13-15mg/Kg UDCA (Active Comparator): Patients will receive standard dosage of 13-15mg/Kg UDCA everyday.
  Interventions: Drug: ursodeoxycholic acid

INTERVENTIONS:
Drug: ursodeoxycholic acid — The two experimental groups will receive reduced dosage of UDCA at 10mg/Kg and 5mg/Kg everyday respectively, while the control group will receive standard dosage of UDCA.The treatment duration will be at least one year.
  Other Names: UDCA

SUMMARY:
This study explores the feasibility of the reducing medication regimen for Ursodeoxycholic Acid(UDCA) in the treatment of primary biliary cholangitis. The participants will be distributed randomly into two experimental groups and one control group. The two experimental groups will receive reduced dosage of UDCA at different level, while the control group will receive standard dosage of UDCA. The effect of therapy will be evaluated every three months.

DETAILED DESCRIPTION:
Primary biliary cholangitis is a chronic, progressive liver disease of autoimmune origin characterized by nonpurulent destruction of intrahepatic ductule, lymphatic infiltration of portal area and long-term intrahepatic cholestasis leading to liver fibrosis and cirrhosis in absence of treatment. The diagnosis is made in the presence of antimitochondrial antibodies (AMA) coupled with an increase in alkaline phosphatase (ALP), a histologic confirmation being mandatory only in seronegative cases or overlap syndrome. Treatment is based on ursodeoxycholic acid (UDCA) and obeticholic acid, which are proved effective in improving biochemical index and preventing disease progression. While obeticholic acid is only approved in USA and Canada, UDCA seem to be the only choice for PBC patients in China. Study has shown that liver function improvement can be expected in six to nine months when patients receive standard dosage( 13 -15mg/kg/d) of UDCA. Recovery of liver function takes two years in 20% of patients ,and five years in 15% to 35% of patients. Lifetime medication is recommended among patients with good respond to UDCA, while the high cost has placed great burden on patients as well as the medical service system. Exploration of the reducing medication regimen of UDCA among stable PBC patients is of great significance under this circumstance. In our study, the 90 recruited PBC patients with a complete response will be distributed randomly into two experimental groups and one control group. The two experimental groups will receive reduced dosage of UDCA at 10mg/Kg and 5mg/Kg respectively, while the control group will receive standard 13-15mg/Kg dosage of UDCA. The effect of therapy will be evaluated every three months, which includes assessment of symptoms, life quality, disease progression, complete blood count, urinalysis, liver biochemical markers (ALT, AST, ALP, GGT, TBIL, DBIL, TP, ALB), blood lipid (CHO, TG, LDL, HDL), immunoglobulins, ESR, AMA, liver morphology and cirrhosis degree, along with peripheral T lymphocyte subpopulations and cytokines test.

ELIGIBILITY:
Inclusion Criteria:

* Satisfied the diagnostic criteria of PBC by the AASLDin 2000;
* Age≥18 years
* Clinical stage 2 and 3 (i.e. abnormal liver function and symptomatic phase);
* Patients with improved liver biochemical index( ALP and AST≤1.5× upper limit of normal, with a normal bilirubin level) after 6 to 12 months treatment of UDCA;
* Informed consent obtained.

Exclusion Criteria:

* Overlapped with other liver diseases (such as HBV, HCV, alcoholic cirrhosis, etc.) or serum ALT, AST more than 2 ULN;
* Decompensation of liver function (Child grade B/C);
* Complicated with important organ failure (such as renal insufficiency), serious infection or other serious complications;
* Pregnancy, preparation for pregnancy or pregnancy Lactation, psychiatric subjects, etc.;
* Participating in other clinical trials or participated in other clinical trials in three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of primary biliary cholangitis | change from baseline to month3,6,9,12.
  Liver biochemical markers (AST and ALP in U/L, TBIL in umol/L) that restored to normal increase(bilirubin>1xULN,ALP≥1.5X ULN, AST≥1.5XULN) again is considered to be PBC recurrence according to the Paris II criteria. The rate of recurrence will be described in percent.

CONTACTS AND LOCATIONS:
Overall Officials: Li Wang, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 6 months after the trial complete
Access Criteria: IPD will be shared by Excel within six months after the trial complete with the public